CLINICAL TRIAL: NCT01387347
Title: A Double-Masked, Randomized, Single-Center Study Evaluating the Safety and Efficacy of 0.1% Tβ4 Ophthalmic Solution Compared to Vehicle on the Signs and Symptoms of Dry Eye in the Controlled Adverse Environment (CAE) Model
Brief Title: Safety and Efficacy of Thymosin Beta 4 Ophthalmic Solution in Patients With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ReGenTree, LLC (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-DE-202
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2012-12

CONDITIONS: Dry Eye Syndrome; Dry Eye
Keywords: Thymosin beta 4; Dry eye syndrome; Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thymosin Beta 4 (Active Comparator): RGN-259 is a preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4
  Interventions: Drug: Thymosin beta 4
- Placebo (Placebo Comparator): The placebo solution is composed of the same excipients as RGN-259 but does not contain Tβ4. The Placebo is identical to the RGN-259 eye drops in color, consistency, and odor.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thymosin beta 4 — A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
  Other Names: Tβ4; RGN-259 (eye drop formulation of Tβ4)
  Arms: Thymosin Beta 4
Drug: Placebo — A preservative-free, sterile eye drop solution containing 0.0% (w/w) Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
  Other Names: Vehicle Control
  Arms: Placebo

SUMMARY:
Thymosin Beta 4 (Tβ4) is a synthetic copy of the naturally-occurring 43-amino acid peptide that is found in a variety of tissues. Tβ4 promotes/accelerates wound repair in dermal, ocular, and cardiac animal models. Two recent pre-clinical evaluations have demonstrated that Tβ4 promotes corneal ocular surface defects healing in animal models of dry eye. RGN-259 (formulation of Tβ4 ophthalmic solution) mechanism of action offers potential to be a product that meets a major unmet medical need in patients with dry eye.

DETAILED DESCRIPTION:
Tβ4 promotes wound repair and regeneration in various tissues. In the eye, it promotes corneal epithelial cell migration, decreases inflammation and has anti-apoptotic activities. It up-regulates the gene expression of laminin-5, a major subepithelial adhesion protein, located in the basement membrane region of the cornea, conjunctiva, and important in wound healing. In compassionate-use cases, Tβ4 has demonstrated efficacy in repairing non-healing neurotrophic corneal ulcers and other corneal epithelial wounds. In twenty-four nonclinical toxicology and safety pharmacology studies, the safety of Tβ4 has been demonstrated for its current and planned uses in man. The results of the two recent dry eye murine mouse model studies show that Tβ4 reduced corneal staining more than positive controls and demonstrated statistically significant reduction in staining compared to vehicle control. The results of these studies, in addition to data from compassionate use studies in patients with non-healing corneal surface defects, suggests that Tβ4 has a significant potential to be an important new safe and effective therapeutic in the treatment of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Have given a written, informed consent.
2. Be able and willing to follow instructions, including participation in study assessments, and be present for the required study visits for the duration of the study.
3. Have a best corrected visual acuity.
4. Have a patient-reported history of dry eye in both eyes.
5. Use and/or desire to use an artificial tear substitute for dry eye symptoms within the past 6 months.
6. A negative urine pregnancy test if female of childbearing potential.
7. Have a corneal fluorescein staining score of ≥ 2 in any corneal surface segment in at least one eye at Visit 1.

   -

Exclusion Criteria:

1. Have contraindications to the use of the study drug.
2. Have known allergy or sensitivity to the study drug or components thereof.
3. Have anterior blepharitis.
4. Be diagnosed with an on-going ocular infection or active ocular inflammation.
5. Use contact lenses within 1 week before Visit 1 or during the course of the study.
6. Have previously had Laser-Assisted in Situ Keratomileusis (LASIK) surgery within 12 months prior to Visit 1.
7. Be currently taking any topical ophthalmic prescription or over-the-counter (OTC) solutions, artificial tears, gels, or scrubs and cannot discontinue these medications for the duration of the trial.
8. Have used topical ocular cyclosporine within 30 days prior to Visit 1.
9. Have had a past or present evidence of malignancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Ora Clinical Research and Development

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at Ora Clinical Research and Development (a medical clinic)by Dr. Gail Torkildsen.The first subject was screened on 13 August 2011 and the last subject last visit to the clinic was on 20 September 2011.
Pre-assignment Details: Subjects who initially qualified for study entry, had adequate baseline staining and redness and positive controlled adverse environment response, were instructed to discontinue all ophthalmic medications and instill a commercially-available sterile irrigating (balanced salt) solution (i.e., the run-in solution) twice a day until Visit 2, Day 0.
Groups:
- Placebo: The placebo solution is composed of the same excipients as RGN-259 but does not contain Tβ4. The Placebo is identical to the RGN-259 eye drops in color, consistency, and odor.
  Placebo : A preservative-free, sterile eye drop solution containing 0.0% (w/w) Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
- Thymosin Beta 4: RGN-259 is a preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4.
  Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
Period: Overall Study
Arm/Group | Placebo | Thymosin Beta 4
Started | 36 | 36
Completed | 34 | 35
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Thymosin Beta 4: RGN-259 is a preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4
  Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Thymosin Beta 4 | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.76) | 57.1 (12.07) | 56.02 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining (Inferior Region) in the Worst Eye in the Controlled Adverse Environment (CAE) Model, Which is a Regulated Environmental Setting Aimed at Exacerbating the Signs and Symptoms of Dry Eye
Description: This is a test that uses orange dye (fluorescein) and a blue light to detect ocular surface defects associated with dry eye. If the test result is normal, the dye remains in the tear film on the surface of the eye and does not adhere to the eye itself. The test is carried out throughout the study till end of treatment Day 29. However, the primary outcome measure itself is determined on Day 29. The scale used to determine the difference in corneal fluorescein staining between RGN-259 and placebo is the ORA scale: 0= no staining (no detectable ocular defect)to 4= confluent staining( severe ocular defect).
  Worst eye: In the case that both eyes were eligible for analysis, the worst eye was chosen as the eye with the greater increase of inferior corneal staining from Visit 1 to Visit 2. If both eyes were equal, the eye with greater ocular discomfort at Visit 2 was chosen as the worst eye. If both eyes were equal at Visit 2, then the right eye was chosen as the worst eye.
Time Frame: Day 29 (end of treatment)
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo is a preservative-free, sterile eye drop solution containing 0% Tβ4 Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0% Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
Arm/Group | Thymosin Beta 4 | Placebo
Number analyzed (Participants) | 36 | 36
units on a scale | 2.08 (0.71) | 1.9 (0.63)
Statistical Analysis 1: Comparison: Thymosin Beta 4 vs Placebo; Inferior corneal fluorescein staining score at Day 29(primary sign) was summarized using descriptive statistics (number of observations, mean, standard deviation, median, minimum, and maximum). Active treatment was compared to placebo using a two-sample t-test assuming unequal variances, assessed at the α = 0.05 level; Test type: Superiority or Other; p = 0.2596, t-test, 2 sided; Mean Difference (Final Values) = 0.18
Statistical Analysis 2: Comparison: Thymosin Beta 4 vs Placebo; Comparison of central corneal fluorescein staining score between the placebo and Thymosin beta 4 groups; Test type: Superiority or Other; p = 0.0075, t-test, 2 sided
Statistical Analysis 3: Comparison: Thymosin Beta 4 vs Placebo; Comparison of superior corneal fluorescein staining score between the placebo and Thymosin beta 4 groups; Test type: Superiority or Other; p = 0.0210, t-test, 2 sided

2. Primary Outcome: Ocular Discomfort in the Worst Eye in the Controlled Adverse Environment(CAE) Model, Which is a Regulated Environmental Setting Aimed at Exacerbating the Signs and Symptoms of Dry Eye.
Description: Dry eye causes ocular discomfort, which is measured using a validated 4-point ORA Scale from the start of the dosing till the end of treatment (Day 29). 0 = no discomfort to 4 = constant discomfort.
  If the measurement is lower, then improvement of ocular discomfort can be inferred. The test is carried out throughout the study till end of treatment Day 29. However, the primary outcome measure itself is determined on Day 29.
  Worst eye: In the case that both eyes were eligible for analysis, the worst eye was chosen as the eye with the greater increase of inferior corneal staining from Visit 1 to Visit 2. If both eyes were equal, the eye with greater ocular discomfort at Visit 2 was chosen as the worst eye. If both eyes had were equal at Visit 2, then the right eye was chosen as the worst eye.
Time Frame: Day 29 (end of treatment)
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Thymosin Beta 4: Thymosin beta 4 solution is a sterile eye drop solution containing 0.1%(w/w) Tβ4. Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, twice a day (BID) for 28 days.
Arm/Group | Placebo | Thymosin Beta 4
Number analyzed (Participants) | 36 | 36
Units on a Scale | 1.3 (1.1) | 1.6 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Thymosin Beta 4; Comparison between the groups uses a two-sample t-test assuming unequal variances, assessed at the alpha = 0.05 level; Test type: Superiority or Other; p = 0.3734, t-test, 2 sided; Mean Difference (Final Values) = 0.3
Statistical Analysis 2: Comparison: Placebo vs Thymosin Beta 4; Comparison of discomfort score between the placebo and Thymosin beta 4 groups on Day 28; Test type: Superiority or Other; p = 0.0244, t-test, 2 sided

3. Secondary Outcome: Number of Adverse Events as a Measure of Safety and Tolerability
Description: The Adverse events, which will be followed, are: impairment of visual acuity, an increase in intraocular pressure (IOP), and an increase in corneal sensitivity in both eyes.
Time Frame: Throughout the study till Day 29
Population: Intention to treat (ITT)
Measure: Number; unit: Events
Groups:
- Placebo: Placebo is a preservative-free, sterile eye drop solution containing 0% Tβ4 (w/w) for direct instillation into each eye twice a day for 29 days.
- Thymosin Beta 4: RGN-259 is a preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye twice a day for 29 days.
Arm/Group | Placebo | Thymosin Beta 4
Number analyzed (Participants) | 36 | 36
Events | 2 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Thymosin Beta 4
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 2/36 | 0/36
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Thymosin Beta 4 (N=36)
General disorder ocular and administration site conditions AND Instillation site pain, (Eye disorders) | 2 (4) | 0 (0) — stinging post administration study gtts (eye drops)

LIMITATIONS AND CAVEATS:
There were no limitations to trial RGN-DE-202 entitled:"Safety and Efficacy of Thymosin beta 4 Ophthalmic Solution in Patients with Dry Eye". All subjects were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less